CLINICAL TRIAL: NCT00379184
Title: Quantitative Assessment of Central Sensitization in Osteoarthritis Patients
Brief Title: Sensitization in Osteoarthritic Knees
Status: Completed | Type: Observational
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: ON-04-014-MBL
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Arthritis
Keywords: arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: Osteoarthritis patients scheduled for Total Knee Arthroplasty.
- B: Osteoarthritis patients not scheduled for Total Knee Arthroplasty.
- C: Healthy volunteers

SUMMARY:
Musculoskeletal pains represent a major part of pain complaints in patients. Moreover, the treatment of musculoskeletal pain conditions by currently available drugs is not optimal (Curatolo and Bogduk 2001). Thus, deep pain is a diagnostic and therapeutic problem, and further insights into the peripheral and central neurophysiologic mechanisms are necessary to improve diagnosis and therapy and to implement a mechanism-based approach. Peripheral sensitization and central hyper excitability are, most likely the important factors for chronic musculoskeletal pain and in particular osteoarthritis (OA).

The focus of this project is to study the involvement of peripheral and central sensitization underlying deep tissue hyperalgesia and referred pain in male and female OA patients.

Adequate quantitative sensory testing assessment techniques for measuring hyper excitability are needed to investigate, in more detail the mechanisms involved in generating the sensitization in OA patients.

DETAILED DESCRIPTION:
Methods

General procedure:

In the Outpatient Department of Clinic Farsoe, Northern Orthopaedic Division patients eligible for participating in the study will be informed and asked to participate. Those who agree and sign the informed consent will be scheduled for the investigational procedures to be performed at the SMI as soon as possible.

At the SMI all patients are interviewed and assessed with the following three procedures with at least 10 minutes between procedures. Duration of visit will be approximately 3 hours in one session.

Procedure 1:

Pressure pain sensitivity and temporal summation of pressure pain

Equipment: computer controlled pressure algometer.

Sites: knee, tibialis anterior, forearm

* Stimulus intensity: pressure pain threshold
* Stimuli number: 10
* Frequency: ISI 1s
* Pain rating: pain intensity, pressure pain threshold, unpleasantness and after-sensations will be collected.

General:

Pressure pain sensitivity and temporal summation of pressure are tested on bilateral knee, tibialis anterior muscle and forearm. Test sites are located and marked according to the landmark stated below. Pressure pain threshold of these test sites are measured first. Sequential stimulations are applied to these test sites respectively to test the pain perception for each press stimulus. Unpleasantness and after-sensations are collected after cessation of sequential stimulation to evaluate the affective aspect of pain.

Specific:

Seven test sites (2 cm proximal to the superior lateral edge of patella, 2 cm proximal to the superior edge of patella, 2 cm proximal to the superior medial edge of patella, 2 cm distal to the inferior lateral edge of patella, 2 cm distal to the inferior medial edge of patella, 5 cm lateral to the superior lateral edge of patella and 5 cm medial to the superior medial edge of patella) are marked around the knee. The site for measuring temporal summation of pain is the most sensitive site among these five sites.

The test site on the arm is 7 cm distal to the lateral humeral epicondyle on the line connecting the lateral epicondyle and the styloid process of the radius, located on the extensor carpi radialis longus muscle.

The test site on the leg is at the tibialis anterior (TA) muscle 14 cm distal to the inferior lateral edge of the patella.

Pressure pain threshold on these test sites are measured. A mechanical pressure stimulus with gradient of 0.3 kg/s will be applied until the subject reports pain and presses a stop button. The PPT measurements start from the contralateral knee of the affected knee.

Sequential stimulation consists of 10 pressure stimuli (1 sec duration) at the pressure pain threshold level. Inter-stimulus interval (ISI) is set to 1 sec. Skin contact between the individual pressure stimuli will be ensured by keeping a constant force of 0.1 kg; i.e. during the series of sequential stimulation the probe has skin contact and is first withdrawn after 10 stimulations. The subjects rate the pain intensity continuously during the sequential stimulation on an electronic visual analogue scale (VAS) on which "0" indicates "no pain" and "10 cm" indicates "maximal pain". Sequential stimulation is to be applied on each test site with at least a 1 min interval. The sequence of test sites is chosen in a randomized way to minimize order effects.

Unpleasantness and after-sensations are collected 15 sec after cessation of sequential stimulation.

Procedure 2:

Referred pain

Equipment: computer controlled pressure algometer, computer-controlled auto-infusion syringe pump.

* Site: tibialis anterior
* Concentration: 6% hypertonic saline.
* Method: continuous infusion.
* Pain rating: pain intensity, pain area drawing (primary and secondary pain area), pressure pain threshold, unpleasantness and after-sensations will be collected.

General:

Hypertonic saline is infused into the tibialis anterior (TA) muscle to elicit local and referred pain. The experiment will be conducted in one leg at a time, by giving a single bolus infusion of hypertonic saline with a time interval of approximately 20 min between each leg. Test sites are located and marked on the TA. Pressure pain thresholds on injection site and front side of ankle are measured before infusion. Hypertonic saline is infused by using a computer-controlled syringe pump. Subjects report pain intensity and draw the pain area induced by infusion. Pressure pain thresholds on injection site and front side of ankle are measured 10 min after infusion- evoked-pain disappears. Unpleasantness and after-sensations for the evoked pain are collected as well.

Specific:

Injection site is placed at the belly of the TA 14 cm distal to the inferior lateral edge of the patella on both legs. At the marked site in the TA a 24G - 40 mm needle will be inserted vertically until a piercing of the muscle fascia is felt, at a depth of approximately 20 mm from the skin surface. Then the plunger of the syringe will be withdrawn to ensure that the needle is deep in the muscle and not in a blood vessel. The needle will then be connected through a polyethylene extension tube (Vygon, France, No. 1155.70) to a 10 ml syringe fitted in a computer-controlled auto-infusion syringe pump (Terumo Terufusion syringe pump, model STC-S27, Type CG). A total volume of 0.5 ml sterile 6% hypertonic saline (58.5 mg/ml, Sygehus Apotekerne, Denmark) will be infused over 20 s into the TA muscle (infusion-rate 90 ml/h).

The pain intensity response is scored on a visual analogue scale (VAS) after the infusion. The subjects mark the painful region(s) on pain maps after the infusion. Local pain is defined as the pain area drawn at the infusion site, referred pain is defined as the pain areas drawn away from the infusion site and radiating pain is defined as the pain areas drawn radiating from the local site into the other regions of the leg.

Pressure pain thresholds on injection site and front side of ankle are measured before and 10 min after infusion when infusion evoked pain disappears.

Unpleasantness and after-sensations for the evoked pain are collected afterwards.

Procedure 3:

Cuff pressure pain and DNIC

Equipment: computer controlled cuff algometer.

* Site: upper arms
* Pain rating: pain intensity, cuff pressure pain threshold, pressure pain threshold, unpleasantness and after-sensations collected.

General:

Continuous cuff pressure stimulation is applied to measure the inhibitory control of the pain sensory system. Cuff stimulation is applied to bilateral upper arms and tibialis anterior (location see procedure 1). Pressure pain threshold on the test sites around knee, on the ipsilateral and contralateral arm (on the belly of biceps brachii) are measured before, during and after cuff pressure stimulation. Cuff pressure stimulation is applied by computer-controlled cuff algometer to induce continuous pain perception for 10 min. Pain intensity of ongoing pain in the stimulated limb and affected knee are rated on electrical VAS.

Specific:

The cuff is wrapped around the middle of both arms. The lower rim of the tourniquet cuff (7.5 cm wide) is at least 3 cm proximal to the cubital fossa. The setup of the cuff algometer is programmed to stop the pressure increase at a preset pain intensity of 4 cm on the VAS and to automatically adjust the pressure to maintain the obtained pain within ±0.5 cm VAS for 10 min or until the subject presses the stop button. If the pain increases over the upper pain limit, the system decreases the pressure until the pain returns into the 'target' zone and vice versa.

When the VAS rise up to 4 cm and keep constant for 1 min, we will measure PPTs on the same test sites except tested arm. Pain intensity of ongoing pain in affected knee and arm which is not stimulated is rated on another electrical VAS during cuff pressure stimulation. Five minutes following deflation, pain intensity of ongoing pain in affected knee and arms is rated. Fifteen minutes following deflation, PPTs are measured on the test sites.

The sequence of test limb is chosen at random to minimize order effects.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis in the knee

Exclusion Criteria:

* No other painful conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with knee OA
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2006-09; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mogens B Laursen, MD, PhD, Principal Investigator — Northern Orthopaedic Division
Locations (1):
- Northern Orthopaedic Division, Clinic Farsoe, Aalborg University Hospital and Aalborg University, Farsø, Northern Jutland, Denmark